CLINICAL TRIAL: NCT06093425
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Study Evaluating Combination of TST001, Pembrolizumab and Chemotherapy as First-Line Treatment in Subjects With Claudin18.2 Positive Locally Advanced or Metastatic Gastric or Gastroesophageal Junction (G/GEJ) Adenocarcinoma
Brief Title: Combination of Osemitamab (TST001), Pembrolizumab and Chemotherapy as First-line Therapy in Advanced or Metastatic GC/GEJ Adenocarcinoma
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Suzhou Transcenta Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: TST001-3001
Record Dates: First submitted 2023-09-24; First posted 2023-10-23 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Gastric Cancer; Gastroesophageal-junction Cancer; Advanced Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — pembrolizumab; Oxaliplatin; Fluorouracil

STUDY DESIGN:
Intervention Model Description: Randomized, Double-Blind, Placebo-Controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- TST001 + PDL-1 + Chemotherapy (Active Comparator): TST001 + Pembrolizumab + Chemotherapy (FOLFOX6 or CapOx)
  Interventions: Drug: Pembrolizumab and either Capcecitabine + Oxaliplatin or Oxaliplatin+Leucovorin + 5-fluorouracil
- Placebo (Placebo Comparator): Placebo + Pembrolizumab + Chemotherapy (FOLFOX6 or CapOx)
  Interventions: Drug: Pembrolizumab and either Capcecitabine + Oxaliplatin or Oxaliplatin+Leucovorin + 5-fluorouracil

INTERVENTIONS:
Drug: Pembrolizumab and either Capcecitabine + Oxaliplatin or Oxaliplatin+Leucovorin + 5-fluorouracil — TST001 will be administered i.v. Q3W along with standard prescribing dose of pembrolizumab Q3W + standard prescribed regimens for FOLFOX6 or CapOx.
  Arms: Placebo
Drug: Pembrolizumab and either Capcecitabine + Oxaliplatin or Oxaliplatin+Leucovorin + 5-fluorouracil — Placebo will be administered i.v. Q3W along with standard prescribing dose of pembrolizumab Q3W + standard prescribed regimens for FOLFOX6 or CapOx.
  Arms: TST001 + PDL-1 + Chemotherapy

SUMMARY:
Gastric/GEJ adenocarcinomas are aggressive tumors with a high probability of death. Current treatment guidelines include two-drug cytotoxic chemotherapy with a fluoropyrimidine (mFOLFOX6: capecitabine or fluorouracil) and a platinum-based agent (CapOx: oxaliplatin or cisplatin). In addition, the FDA has approved nivolumab, a PD-1 checkpoint inhibitor, in combination with chemotherapy as first line treatment for advanced or metastatic gastric/GEJ cancer. TST001 is a recombinant humanized monoclonal antibody against Claudin 18.2 (a tumor marker found in gastric/GEJ cancer. In this study, the combination therapy of chemotherapy or chemotherapy and pembrolizumab with and without TST001 could provide additional benefits to the management of these tumors.

DETAILED DESCRIPTION:
This Phase 3, randomized, double-blind, placebo-controlled study is designed to evaluate the safety and efficacy of TST001 in combination with pembrolizumab and chemotherapy or chemotherapy alone in subjects with tumors that express markers (HER2 negative, Claudin18.2 positive, known PD-L1 CPS status) in locally advanced or metastatic gastric/GEJ adenocarcinoma. Patients will be randomized in a 1:1 ration to receive TST001 or placebo in combination with nivolumab and chemotherapy or with chemotherapy alone.

ELIGIBILITY:
Inclusion Criteria:

* 1. ≥18 years of age on day of signing informed consent. 2. Histologically or cytologically confirmed diagnosis of previously untreated, unresectable locally advanced or metastatic G/GEJ adenocarcinoma.

  3. Must be willing and able to provide archival or fresh tissue sample, a formalin-fixed, paraffin-embedded (FFPE) block, or 151 or more unstained, freshly cut, serial sections (on slides) from an FFPE tumor specimen or fresh biopsy tissue from a tumor lesion (either primary or metastatic) not previously irradiated fixed in formalin solution. FFPE tissue blocks are preferred to slides. Notes: details pertaining to tumor tissue submission can be found in the Laboratory Manual. Fresh biopsies are not required for study entry and will not be covered as part of the study procedures. Handling of the fresh biopsy tissue is an alternative offered to investigators in case they plan to biopsy the subjects as part of their standard of care; the fresh sample can be sent directly to the central laboratory if it is more convenient to the sites.

  4. Positive CLDN18.2 expression in tumor tissue confirmed by the central laboratory at screening using CTA (Claudin 18.2 IHC 14G11 pharmDx).

  5. Must have at least one measurable lesion or evaluable disease by CT or MRI per RECIST 1.1 criteria as assessed locally by the investigator; radiographic tumor assessment should be performed within 28 days prior to randomization.

  6. Subjects should be eligible to receive chemotherapy and pembrolizumab per the investigator judgement.

  7. Known PD-L1 CPS Status (tested by central laboratory to provide CPS status by PD-L1 IHC 22C3 pharmDx).

  8. Have an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1 assessed within 14 days before randomization.

  9. Subjects who have AEs due to previous anticancer therapies must have recovered to ≤Grade 1 or pre-treatment status. Subjects with endocrine-related AEs who are adequately treated with hormone replacement or subjects who have ≤Grade 2 neuropathy are eligible.

  10. Have a life expectancy of greater than 12 weeks. 11. Demonstrate adequate organ function.

Exclusion Criteria

1. Has received any prior systemic anticancer treatment (chemotherapy, immunotherapy, biologic therapy, or targeted therapy) for G/GEJ adenocarcinoma. Neo/adjuvant treatment is permitted as long as it was completed at least 6 months prior to randomization.
2. Has received prior radiotherapy within 2 weeks before randomization; Note: Subjects must have recovered from all radiation-related toxicities. A previously irradiated lesion can be used as measurable lesion as long as it progressed post radiation therapy.
3. Has received anti-CLDN18.2 agents at any time.
4. Has received any traditional Chinese medicine or proprietary Chinese medicine with anti-tumor effect within 7 days before randomization.
5. Has received vaccines (live, attenuated, or research vaccines) within 30 days before randomization. Administration of killed vaccines is allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 820 (Estimated)
Dates: Start 2026-06-30 (Estimated); Primary Completion 2029-10-01 (Estimated); Study Completion 2030-01-31 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) based on RECIST (v1.1) | Date of randomization until the date of documented progression or date of death due to any cause, whichever comes first up to 24 months after last dose.
  Compare PFS of patients treated with TST001 or Placebo in combination with pembrolizumab and chemotherapy

SECONDARY OUTCOMES:
Overall Survival (OS) based on RESIST | Time from date of randomization until the date of death due to any cause, assessed up to 24 months after last dose.
  Compare OS of patients treated with TST001 or Placebo in addition to CapOx or mFOLFOX6 and pembrolizumab or CapOx or mFOLFOX6
Overall Response Rate (ORR) based on RESIST (v1.1) | Date of randomization up to 24 months after last dose
  Compare OOR patients treated with TST001 or Placebo in addition to CapOx or mFOLFOX6 and pembrolizumab or CapOx or mFOLFOX6.
Quality of Life (QOL) assessed on EuroQol EQ5D-5L | Date of randomization until the date of documented progression, assessed up to 24 months after last dose
  Change in QOL assessments from baseline of patients treated with TST001 or Placebo in addition to mFOLFOX6 and pembrolizumab or CapOx or mFOLFOX6. Assessments include Cancer QOL questionnaires (QLC-STO22, EQ5D-5L, and QLQ-C30)
Disease Control Rate (DCR) based on RESIST assessed as the percentage of subjects with measurable disease | Date of randomization up to 24 months after last dose
  Compare DCR of patients treated with TST001 or Placebo in addition to CapOx or mFOLFOX6 and pembrolizumab or CapOx or mFOLFOX6.
Duration of Response (DOR) based on RESIST (log-rank test) | From date of randomization up to 24 months after last dose
  Compare DOR of patients treated with TST001 or Placebo in addition to CapOx or mFOLFOX6 and pembrolizumab or CapOx or mFOLFOX6.
Time to Response (TTR) based on RESIST | Date of randomization up to 24 months after last dose
  Compare TTR of patients treated with TST001 or Placebo in addition to CapOx or mFOLFOX6 and pembrolizumab or CapOx or mFOLFOX6 based on CR or PR.

IPD SHARING:
Plan to Share IPD: No
Summary of study results will be available through Clinicaltrials.gov